CLINICAL TRIAL: NCT07169617
Title: Evaluating the Feasibility of a Survivin Peptide Vaccine (SurVaxM) as an Interception Agent in Patients at High Risk for Lung Cancer
Brief Title: Testing the SurVaxM Vaccine for Lung Cancer Prevention
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2025-06377; NCI-2025-06377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI24-19-01 (Other: Northwestern University); NWU24-19-01 (Other: DCP); P30CA060553 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; montanide ISA 51; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (SurVaxM, montanide, sargramostim) (Experimental): Patients receive SurVaxM with montanide SC followed by sargramostim SC on day 0, week 2, week 4, and week 6. Patients then receive a booster dose of SurVaxM with montanide SC followed by sargramostim SC on week 18. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Montanide ISA 51 VG; Other: Questionnaire Administration; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Montanide ISA 51 VG — Given SC
Other: Questionnaire Administration — Ancillary studies
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: SVN53-67/M57-KLH Peptide Vaccine — Given SC
  Other Names: SurVaxM

SUMMARY:
This phase II trial tests how well a survivin peptide vaccine called SurVaxM works in preventing lung cancer in high risk patients. Upon administration, the SurVaxM vaccine activates the immune system to produce an immune cell response against cancer cells that express a protein called survivin. This may result in decreased tumor cell proliferation and lead to tumor cell death. SurVaxM is given with montanide, a substance that helps the immune system respond to the SurVaxM vaccine, followed by sargramostim, which is given to increase the number of white blood cells in the body. The SurVaxM vaccine may help the body make special proteins called antibodies, which may be helpful in preventing the development of lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of SVN53-67/M57-KLH peptide vaccine (SurVaxM) administration on the generation of a systemic anti-survivin immune response.

SECONDARY OBJECTIVES:

I. To assess the proportion of participants needing a 3-month booster dose to achieve seroconversion.

II. To assess the proportion of participants mounting a cellular immune response to SurVaxM vaccination.

III. To assess the safety profile of SurVaxM administration in this population.

EXPLORATORY OBJECTIVES:

I. To associate participants' demographic and clinical characteristics with outcomes (seroconversion or needing the 3-month booster).

II. Correlation of human leukocyte antigen (HLA) typing and the association of HLA types to humoral and/or cellular responses.

OUTLINE:

Patients receive SurVaxM with montanide ISA 51 VG (montanide) subcutaneously (SC) followed by sargramostim SC on day 0, week 2, week 4, and week 6. Patients then receive a booster dose of SurVaxM with montanide SC followed by sargramostim SC on week 18. Patients also undergo collection of blood samples throughout the trial.

After completion of study intervention, patients are followed up at weeks 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Former and current smokers (male and female) with a >= 20 pack year smoking history
* Prostate, Lung, Colorectal and Ovarian (PLCO)m2012 Lung Cancer Risk Prediction Score > 1.34%
* Participants >= 18 years old will be enrolled. Because no dosing or adverse event (AE) data are currently available on the use of SurVaxM in participants < 18 years of age, children and adolescents are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 60%)
* Platelets >= 100,000/microliter
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)

  * Note: Higher total bilirubin levels (=< 3 mg/dL) can be allowed if due to known benign liver condition, i.e. Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Serum creatinine =< 1.5 x institutional upper limit of normal
* The effects of SurVaxM plus montanide on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of autoimmune disease necessitating systemic immunosuppression, immunodeficiency, and/or organ allograft
* Participants may not be receiving any other chemotherapy (except hormonal agents), immunotherapy or investigational agent, or any immunosuppressive agent, including systemic steroids, including those given after organ transplant
* Participants with current or prior malignancy except for the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years before screening and felt to be at low risk for recurrence by treating physician
  * Adequately treated carcinoma-in-situ or basal cell carcinoma of the skin without current evidence of disease
  * Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanomatous skin cancer
  * Prior or current malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen (e.g., localized prostate cancer) may be included
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to montanide or granulocyte-macrophage colony-stimulating factor (GM-CSF)
* Uncontrolled intercurrent illness, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because of the unknown effects of SurVaxM plus montanide on the fetus. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with SurVaxM plus montanide, breastfeeding should be discontinued if the mother is treated with SurVaxM plus montanide
* Individuals participating in another interception trial with an immunomodulatory agent will be excluded from participation in this trial for a washout period of 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | Up to week 20
  Seroconversion rate will be summarized as the frequency and proportion of participants who achieved sufficient seroconversion, which will be reported with the corresponding 95% confidence intervals. A one-sample exact test for one proportion will be used to test whether seroconversion rate exceeds the unacceptably low rate of 50%.

SECONDARY OUTCOMES:
Proportion of participants who require a 3-month booster to achieve seroconversion | At week 18
  Proportions will be reported with the corresponding confidence intervals.
Proportion of participants who achieve seroconversion | By 3 months
  Proportions will be reported with the corresponding confidence intervals.
Proportion of participants who do not achieve seroconversion at 3 months but achieve seroconversion 2-4 weeks after receiving a 3-month booster | Up to week 20
  Proportions will be reported with the corresponding confidence intervals.
Proportion of participants who do not achieve seroconversion | Up to week 20
  Proportions will be reported with the corresponding confidence intervals.
Cellular responses to the administration of SVN53-67/M57-KLH peptide vaccine | Before the administration of the first dose, 2-4 weeks after completion of the four priming doses, prior to receiving the booster, and 2-4 weeks after completion of the booster
  Will be measured on peripheral blood mononuclear cells. Will tabulate the proportion of participants mounting a cellular response using flow cytometry.
Incidence of adverse events | Up to week 24
  Participants will also be provided with a participant diary, thermometer, and injection site reaction measuring tools to assist in collection and documentation of adverse events post-injection. All adverse events attributable to the vaccine as well as their severity will be reported in a descriptive format. The incidence rate and severity of each attributable adverse event will be tabulated and reported. Adverse events will be assessed using Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Seroconversion rate | Up to week 20
  Will perform exploratory analyses associating participants' demographic and clinical characteristics with outcomes using Wilcoxon ranksum tests to compare continuous variables between responders and non-responders using Fisher's exact test or chi-squared test to compare categorical variables between responders and non-responders. Multivariable logistic regression models will be used to examine the effects of multiple risk factors simultaneously.
Proportion of participants who require a 3-month booster to achieve seroconversion | At week 18
  Will perform exploratory analyses associating participants' demographic and clinical characteristics with outcomes using Wilcoxon ranksum tests to compare continuous variables between responders and non-responders using Fisher's exact test or chi-squared test to compare categorical variables between responders and non-responders. Multivariable logistic regression models will be used to examine the effects of multiple risk factors simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Saikrishna S Yendamuri, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Tennessee - Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm